CLINICAL TRIAL: NCT05012254
Title: Nivolumab Plus Ipilimumab Plus Two Cycles of Platinum-based Chemotherapy as First Line Treatment for Stage IV/Recurrent Non-small Cell Lung Cancer (NSCLC) Patients With Synchronous Brain Metastases
Brief Title: Nivolumab and Ipilimumab Plus Chemotherapy for Patients With Stage IV Lung Cancer With Brain Metastases
Acronym: NIVIPI-Brain
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 21/02_NIVIPI-Brain; 2021-000425-27 (EudraCT Number)
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Brain Metastases, Adult; Lung Cancer
Keywords: Lung Diseases; Chemotherapy; Immunotherapy; Induction chemotherapy; Maintenance treatment; Nivolumab; Ipilimumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Lung Neoplasms; Lung Diseases | interventions — Ipilimumab; Nivolumab; Carboplatin; Cisplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Induction treatment + Maintenance (Experimental): Induction: 2 cycles of platinum-based chemotherapy plus (Nivolumab + Ipilimumab):
  - Non-squamous NSCLC patients: Pemetrexed: 500 mg/m2 IV, Q3W Carboplatin: AUC 5 o 6 or Cisplatin: 75 mg/m2 IV, Q3W Nivolumab: 360 mg IV Q3W Ipilimumab: 1mg/kg IV Q6W
  2 cycles will be administered at 21-day intervals (Q3W) for Pemetrexed, Carboplatin/Cisplatin and Nivolumab. Ipilimumab will be administered at 42 days interval (Q6W).
  - Squamous NSCLC patients: Paclitaxel: 200 mg/m2 IV, Q3W Carboplatin: AUC 5 o 6, Q3W Nivolumab: 360 mg IV, Q3W Ipilimumab: 1mg/kg IV, Q6W
  Maintenance: following two cycles of chemo-immunotherapy the patients will receive:
  Nivolumab: 360 mg IV, Q3W Ipilimumab: 1mg/kg IV, Q6W
  Immunotherapy will be administered until disease progression, unacceptable toxicity, loss of clinical benefit or up to a maximum of 2 years of treatment.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Ipilimumab — Patients will receive Ipilimumab 1mg/Kg administered by IV infusion every 42 days (Q6W) until disease progression, unacceptable toxicity, loss of clinical benefit as judged by the investigator or up to a maximum of 2 years of treatment.
  Structure: is a fully human monoclonal antibody with two heavy chains and two kappa light chains linked together by way of disulfide bonds. The molecular weight is approximately 148 kDa and it exists in solution at a physiologic pH of 7.0.
  Route of administration: Intravenous infusion.
  Other Names: Yervoy
Drug: Nivolumab — Patients will receive Nivolumab 360 mg administered by IV infusion every 21 days (Q3W) until disease progression, unacceptable toxicity, loss of clinical benefit as judged by the investigator or up to a maximum of 2 years of treatment.
  Structure: Nivolumab is a soluble protein consisting of 4 polypeptide chains, which include 2 identical heavy chains and 2 identical light chains.
  Route of administration: Intravenous infusion.
  Other Names: Opdivo
Drug: Carboplatin — Patients will receive Carboplatin AUC 5 or 6 administered by IV infusion every 21 days (Q3W), for 2 cycles.
  Structure: The cis-diamino (cyclobutane-1, 1 dicarboxylate) platin. Stability: 24 hours at ambient temperature in 5% glucose, glucosa or physiologic saline. It is recommended not to dilute with chlorinated solutions since this could affect the carboplatin.
  Route of administration: Intravenous infusion. Guidelines of Carboplatin administration: According to the standard of each center.
  Other Names: Paraplatin
Drug: Cisplatin — Patients will receive Cisplatin 75mg/m2 administered by IV infusion every 21 days (Q3W), for 2 cycles.
  Structure: (CAS No. 15663-27-1, MF-Cl2H6N2Pt; NCF-119875), cisplatinum, also called cis-diamminedichloroplatinum(II), is a metallic (platinum) coordination compound with a square planar geometry. It is a white or deep yellow to yellow-orange crystalline powder at room temperature.
  Stability: Do not store above 25°C. Do not refrigerate or freeze. Keep container in the outer carton to protect from light. Following dilution in 0.9% sodium chloride injection, chemical and physical in-use stability has been demonstrated for up to 14 days at 20°C.
  Route of administration: Intravenous infusion. Guidelines of Cisplatin administration: According to the standard of each center.
  Other Names: Cis-diamminedichloroplatinum; Platinol
Drug: Paclitaxel — Patients will receive Paclitaxel 200mg/m2 administered by IV infusion every 21 days (Q3W), for 2 cycles.
  Structure: A diterpene whose composition is: 5b, 20-epoxy-1, 2a, 4,7b, 10b, 13a-hexahidroxytax-11-en 9 one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)- N-benzoyl-3-phenylisoserine.
  Stability: Concentrations of 0.3-1.2 mg/ml in 5% dextrose or normal saline have demonstrated chemical and physical stability for more that 27 hours at ambient temperature (25ºC approximately). The intact vial must be stored between 15º and 25ºC.
  Guidelines of Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol
Drug: Pemetrexed — Patients will receive Pemetrexed 500mg/m2 administered by IV infusion every 21 days (Q3W), for 2 cycles.
  Structure: Pemetrexed disodium (ALIMTA®, pemetrexed) is a novel pyrrol [2,3 d]-pyrimidine based folic acid analogue.
  Route of administration: Intravenous infusion. Guidelines of Pemetrexed administration: According to the standard of each center
  Other Names: Pemetrexed disodium; ALIMTA

SUMMARY:
This is an open-label, non-randomised, phase II, multicenter clinical trial.

71 stage IV or recurrent, non-small cell lung cancer patients with synchronous brain metastases will be enrolled in this trial to evaluate the efficacy of Nivolumab plus Ipilimumab plus two cycles of platinum-based chemotherapy as first line treatment.

DETAILED DESCRIPTION:
This is an open-label, non-randomised, phase II, multicenter clinical trial. The total sample size is 71 patients. The population to be included are stage IV or recurrent, non-small cell lung cancer patients with synchronous brain metastases.

Patients randomised will receive induction treatment with two cycles of platinum-based chemotherapy plus Nivolumab and Ipilimumab. At the end of induction treatment the patient with start maintenance with Nivolumab and Ipilimumab until disease progression, unacceptable toxicity, loss of clinical benefit as judged by the investigator or up to a maximum of 2 years of treatment

The primary objective of this trial is to determine the rate of intracranial clinical benefit, defined as the percentage of patients who had lack of radiological or clinical progression for at least 6 months according to RANO-BM assessment criteria.

Patient accrual is expected to be completed within 1.5 years, treatment is planned to extend for 1 year and the patients will be followed up for 2 years. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* COHORT A Patients with histologically or cytologically confirmed stage IV NSCLC who did not receive any prior systemic therapy for advanced disease and have synchronous untreated brain metastases which does not cause neurologic symptoms and does not require systemic corticosteroid treatment within 10 days before initiating study treatment (controlled seizures with antiepileptic drugs should be allowed).
* COHORT B Patients with histologically or cytologically confirmed stage IV NSCLC who did not receive any prior systemic therapy for advanced disease and have synchronous brain metastasis causing neurologic signs and symptoms controlled with medium-low doses of corticosteroids (≤ 25mg/d of prednisone or ≤ 4mg/d of dexamethasone) but have good performance status (ECOG PS0-1). At least one untreated brain lesion in patients who already received focal radiotherapy (stereotactic focal radiotherapy) of prior brain lesions are eligible if novel brain lesions appear which are measurable and not suitable for focal radiotherapy.3. Patients with early or locally advanced NSCLC who have recurred after 6 months of completing adjuvant or neoadjuvant chemotherapy and have brain metastases are also eligible
* ECOG performance status 0-1
* Patients aged ≥ 18 years
* Systemic measurable disease by computed tomography (CT) per response evaluation criteria in solid tumors version (RECIST) 1.1 criteria and brain measurable disease by magnetic resonance imaging (MRI) per RANO-BM criteria.
* Availability of a formalin-fixed paraffin-embedded block containing tumor tissue or 10 unstained slides. Archival tumor tissue can be sent if it was obtained less than 12 months ago.
* Correct hematological, hepatic and renal function. i. Neutrophils ≥ 1500×109/L ii. Platelets ≥ 100 ×109/L iii. Hemoglobin ≥ 9.0 g/dL iv. Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 45 mL/min (if using the Cockcroft-Gault formula below): a. Female CrCl = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL b. Male CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL v. AST/ALT ≤ 3 x ULN. Patients with documented liver metastases: AST and/or ALT ≤ 5 × ULN vi. Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 x ULN) vii. PT/APTT ≤ 1.5 × upper limit of normal (ULN). This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose
* Patient consent must be obtained in the appropriate manner as established in the applicable local and regulatory requirements
* Patients must be accessible for treatment and follow-up
* Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 3 days before randomization.
* All sexually active men and women of childbearing potential must use a highly effective contraceptive method (<1% failure rate) during the study treatment and for a period of at least 5 months for females and 7 months for males following the last administration of trial drugs.

Exclusion Criteria:

* Patients with a history of other malignant diseases within the past 3 years, with the exception of the following:

  * properly treated non-melanotic skin cancer
  * cancer in situ treated with curative intent
  * nonmuscular propria invasive carcinoma of the bladder
  * or other malignancies treated with curative intent and without signs of disease for a period of > 3 years after the end of the treatment and which, in the opinion of the physician in charge of their treatment, do not present a substantial risk of relapse of the previous malignant disease.
* Patients harboring epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) and ROS Proto-Oncogene 1 (ROS1) rearrangements sensitive to available targeted inhibitor therapy
* Patients with a combination of small cell lung cancer and non-small cell lung cancer, a carcinoid lung tumor or large cell neuroendocrine carcinoma
* Patients that received live attenuated vaccines within 30 days prior to randomization
* Leptomeningeal carcinomatosis or metastases in the brain stem, mid-brain, pons, medulla or causing obstructive hydrocephalus
* Single exclusive brain metastasis amenable to surgical treatment or radiosurgery
* Prior surgical resection of brain or spinal lesions in the prior 28 days
* Patients who have received prior neoadjuvant, adjuvant chemotherapy, radiotherapy, or chemo-radiotherapy with curative intent for non-metastatic disease less than 6 months before enrollment since the last chemotherapy, radiotherapy, or chemo-radiotherapy
* History of a primary immunodeficiency, history of organ allogeneic transplantation, use of immunosuppressive drugs within 28 days before randomization or previous history of toxicity of severe immune mechanism (grade 3 or 4) with other immunological treatments
* Patients with an active, known or suspected autoimmune disease. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to be enrolled
* Patients with active or uncontrolled infections or with serious medical conditions or disorders that may not allow patient management as established in the protocol
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of radiation pneumonitis put of the radiation field on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Significant comorbidities that preclude the administration of chemotherapy according to the investigator's criteria
* Any positive test result for hepatitis B virus or hepatitis C virus indicating presence of virus, e.g. Hepatitis B surface antigen (HBsAg, Australia antigen) positive, or Hepatitis C antibody (anti-HCV) positive (except if HCV-RNA negative)
* Previous treatment with immune checkpoint inhibitors
* Patients who have suffered untreated and / or uncontrolled cardiovascular disorders and / or who have symptomatic cardiac dysfunction (unstable angina, congestive heart failure, myocardial infarction in the previous year or ventricular cardiac arrhythmias that require medication, history of atrioventricular conduction of second or third degree)
* Pregnant or breastfeeding women
* History of allergy or hypersensitivity to any of the study drug components
* Patients with a condition other than brain metastases requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Rate of intracranial clinical benefit | From the date of the end of treatment until the date of last follow up, assessed up to 24 months
  Defined as the percentage of patients who had lack of radiological or clinical progression for at least 6 months according to RANO-BM assessment criteria

SECONDARY OUTCOMES:
To assess the efficacy of the treatment in terms of the Progression Free Survival (PFS) | From the date of the end of treatment until the date of last follow up, assessed up to 24 months
  PFS defined as systemic PFS (excluding CNS) as per RECIST version 1.1 and PFS in the CNS as per RANO-BM criteria
To evaluate the Overall Response Rate (ORR) of the treatment | From the date of the end of treatment until the date of last follow up, assessed up to 24 months
  Intracranial ORR, defined as a complete response or partial response as determined by the investigator according to RANO for brain disease. Systemic ORR, defined as a complete response or partial response as determined by the investigator according to RECIST v1.1. criteria for systemic disease.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 100 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Nadal, MD, Principal Investigator — Fundación GECP Investigator
Locations (18):
- Spain (18):
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Provincial de Castellón, Castellon, Castellon
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario de León, León
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital 12 De Octubre, Madrid
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitari Son Llatzer, Palma de Mallorca
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org